CLINICAL TRIAL: NCT04008914
Title: Readmission Risk Factors and Heart Failure With Preserved Ejection Fraction
Status: Completed | Type: Observational
Sponsor: Ascension Macomb-Oakland Hospital (Other)
Responsible Party: Principal Investigator, Dustin Harmon, Principle Investigator, Ascension Macomb-Oakland Hospital
Other Study IDs: AscensionMacombOaklandH
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure; Preserved Ejection Fraction
Keywords: Heart Failure; Readmission Risks
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- readmission at 30 days
  Interventions: Other: retrospective observation
- readmission at 90 days
  Interventions: Other: retrospective observation

INTERVENTIONS:
Other: retrospective observation — Retrospective review of study patients excluded from the CONNECT- HF trial who were discharged with a diagnosis of HFpEF between August 1, 2017 and March 1, 2018. Readmission rate at 30 and 90 days along with patient demographics and associated comorbidities were analyzed.

SUMMARY:
Retrospective review of 492 patient from a small community hospital who did not qualify for participation in the Connect HF study sponsored by DCRI.

DETAILED DESCRIPTION:
Retrospective review of adults above the age of 18 with a primary diagnosis of HFpEF between August 2017 and March 2018. Subjects had to fall into one of two classifications (NYHA Class II-IV or ACC/AHA Stage B-D) and had a life expectancy greater than 6 months are included. Individuals with a terminal illness other than HF, prior heart transplant or on a transplant list, or current/ planned left ventricular assist device excluded. The primary objective of this study is to identify risk factors for readmission in patients discharged with a diagnosis of HFpEF.

ELIGIBILITY:
Inclusion Criteria:

* History of Heart failure diagnosis admitted for treatment
* Ejection fraction < 40% by echocardiogram

Exclusion Criteria:

* Ejection fraction >40% by echocardiogram
* Chronic Kidney disease requiring dialysis
* Terminal illness
* New onset diagnosis of Heart Failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All
Sampling Method: Non-Probability Sample
Enrollment: 492 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
Readmission Risk Factors and Heart Failure with Preserved Ejection Fraction | August 1, 2017 though March 1, 2018
  Retrospective review to identify risk factors for readmission in patients discharged with a diagnosis of HFpEF.

CONTACTS AND LOCATIONS:
Overall Officials: Dustin Harmon, DO, Principal Investigator — Ascension Macomb-Oakland Hospital
Locations (1):
- Ascension Macomb-Oakland Hospital, Warren, Michigan, United States